CLINICAL TRIAL: NCT04882306
Title: The ABC Study: Assessment of Breast Density Classification Via Algorithm Development Using Microwave Imaging in Breast Clinics
Brief Title: The ABC Study: Assessment of Breast Density Classification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Micrima, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTOCOL-P2-054
Record Dates: First submitted 2021-03-19; First posted 2021-05-11 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study group (Other)
  Interventions: Device: Bilateral MARIA scan

INTERVENTIONS:
Device: Bilateral MARIA scan — After consent has been given, the participant's breast will be fitted by the operator using a clear plastic cup to determine their corresponding MARIA® cup insert size. Once this has been determined, participants will be required to lie prone with their breast pendent through an aperture in the MARIA® patient bed. The cup insert will contain a layer of coupling fluid. The hemispherical cup inserts, and array are brought into contact with the breast. Depending on the patient's breast size, one or more cup inserts may be placed in the array to ensure a good but non-compressing fit between the breast and the system interface. The scan sequence will then be performed, this takes a couple of minutes.

SUMMARY:
The MARIA® breast imaging system is a CE-marked radiofrequency (RF) medical imaging device. The system employs an electromagnetic imaging technique that exploits the dielectric contrast between normal and cancerous tissues. It is the intention that MARIA® will be able to offer a breast density classifier to clinician's but for this project to be successful, data is required. This study will collect the data required for the classifier to be developed.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a subject must meet all the following criteria:

  * Attending a symptomatic or assessment breast clinic at the study site
  * Female sex
  * 18 years or older
  * Able to provide informed consent
  * Not in any identified, vulnerable group

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:

  * Unable to mount MARIA® patient bed
  * Unable to lie in the prone position for a period of up to 15 minutes
  * Patients who have undergone biopsy less than 5 days before the MARIA® scan
  * Patients with implanted electronics
  * Patients with breast implants
  * Patients with nipple piercings (unless they are removed prior to the MARIA® scan)
  * Breast sizes too small or too large to be suitable for the array

Participants recruited the same day are not subject to any additional screening criteria other than that described above. However, participants being recruited and consenting to the use of previously- taken mammography will need to provide information on key points in order to assess the eligibility of their mammograms for use. This will include information on:

* Whether they have initiated or discontinued use of a hormonal contraceptive since their last mammogram
* Whether they have initiated or discontinued use of hormone replacement therapy since their last mammogram
* Whether they believe that they have had a change in menopausal status since their last mammogram Participants who answer yes to any of the above will not be eligible for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
The creation of the required dataset to develop the breast density classification algorithm | 12 months
  Dataset of information containing ground truth breast density from mammogram
The creation of that algorithm | 12 months
  Using the current breast density algorithm developed for MARIA to analyse the MARIA images and compare that to the mammographic ground truth
The assessment of the performance of that algorithm to measure breast density when compared to the ground truth of the Boyd score | 12 months
  Analyse the values obtained from both the MARIA algorithm and the mammographic ground truth, and look for correlation using the Boyd percentage score of breast density.

SECONDARY OUTCOMES:
Understand participant acceptability of the MARIA® scan | 12 months
  Using a specially-designed patient questionnaire, analyse feedback on the MARIA scan experience using a scale from Very acceptable-Acceptable-Neither acceptable or unacceptable-Unacceptable-Very unacceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- North Devon Breast Screening Service- In Health, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No